CLINICAL TRIAL: NCT06221930
Title: Researching the Effectiveness of Attexis, a Digital Health Application for Adults With Attention Deficit Hyperactivity Disorder - a Randomized Controlled Trial
Brief Title: Researching the Effectiveness of Attexis, a Digital Health Application for Adults With Attention Deficit Hyperactivity Disorder
Acronym: READ-ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaia AG (Industry)
Collaborators: Zentrum für Integrative Psychiatrie Kiel (Unknown); University Hospital, Saarland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: attexis RCT 2024
Record Dates: First submitted 2024-01-15; First posted 2024-01-24 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Adult Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- attexis + TAU (Experimental): Participants allocated to the intervention group will receive access to attexis in addition to treatment as usual (TAU).
  attexis is a digital health application designed for individuals with adult attention deficit hyperactivity disorder (ADHD), accessible through a web browser. The application focuses on treatment methods derived from cognitive behavioral therapy (CBT). Topics addressed by attexis are attention, self-image, impulsivity and physical exercise, problem-solving strategies, and resources.
  The program operates through interactive "dialogues", which are accompanied by illustrations, audio recordings, motivational text messages, worksheets, and summaries. Users are also encouraged to regularly complete short questionnaires to monitor their complaints. Once registered, the program remains accessible for 180 days.
  Interventions: Behavioral: attexis
- TAU (No Intervention): Participants allocated to the control group will receive access to treatment as usual (TAU).

INTERVENTIONS:
Behavioral: attexis — Participants will receive access to the digital health intervention attexis in addition to TAU.
  Arms: attexis + TAU

SUMMARY:
In this randomized controlled clinical trial, 326 patients with ADHD will be investigated regarding the effectiveness of a digital therapeutic for improved ADHD symptomatology, the unguided online intervention attexis. Inclusion criteria are: male, female or non-binary, age 18-65, diagnosis of ADHD, elevated levels of ADHD symptoms (score of ≥17 either on the inattention subscale or on the impulsivity/hyperactivity subscale of the ASRS v1.1), stable treatment for at least 30 days at time of inclusion, sufficient German skills, and consent to participation. Exclusion criteria are: Diagnosis of any other severe psychiatric disorder and plans to change treatment in the upcoming three months. Patients will be randomized and allocated to either an intervention group, receiving access to attexis in addition to TAU, or a control group, receiving access to TAU only. Primary endpoint will be self-rated ADHD symptomatology, assessed via the ASRS v1.1, with three months post-allocation being the primary time point for assessment of effectiveness. Six months post allocation will be used as a timepoint for follow-up assessment of endpoints. Secondary endpoints will be depressive symptoms, self-esteem, work and social functioning, and health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* women, men, non-binary
* age 18-65 years
* diagnosis of ADHD (assessed via DIVA)
* ADHD severity score (cut-off): score of ≥17 either on the inattention subscale or on the impulsivity/hyperactivity subscale of the ASRS v1.1
* stable treatment (psychotherapy, medication, no treatment, …) for at least 30 days at the time of inclusion
* consent to participation
* sufficient knowledge of the German language

Exclusion Criteria:

* diagnosis of another severe psychiatric disorder (severe affective disorder, autism spectrum disorder, psychotic disorder, Borderline personality disorder, antisocial personality disorder, substance use disorder, suicidality)
* plans to change treatment (psychotherapy, medication, …) in the upcoming three months after inclusion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 337 (Actual)
Dates: Start 2024-03-11 (Actual); Primary Completion 2024-09-25 (Actual); Study Completion 2024-12-25 (Actual)

PRIMARY OUTCOMES:
ADHD Symptom Severity | 3 months
  ASRS v1.1. Total score ranging from 0-72; higher scores mean more ADHD symptoms (worse outcome).

SECONDARY OUTCOMES:
Depressive Symptomatology | 3 months, 6 months
  PHQ-9. Total score ranging from 0-27; higher scores mean more depressive symptomatology (worse outcome).
Self Esteem | 3 months, 6 months
  Rosenberg Self Esteem Scale (RSES). Total score ranging from 0-30; higher scores mean higher self-esteem (better outcome).
Functioning | 3 months, 6 months
  Work and Social Adjustment Scale (WSAS). Total score ranging from 0-40; higher scores mean higher impairment (worse outcome).
Health-Related Quality of Life | 3 months, 6 months
  AQoL-8D. Total score ranging from 0-100; higher scores mean higher quality of life (better outcome).
ADHD Symptom Severity | 6 months
  ASRS v1.1. Total score ranging from 0-72; higher scores mean more ADHD symptoms (worse outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Eva Fassbinder, MD, Principal Investigator — Zentrum für Integrative Psychiatrie Kiel
Locations (1):
- GAIA AG, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No